CLINICAL TRIAL: NCT02351895
Title: Effect of Copper Impregnated Textiles on Healthcare Associated Infections and Antibiotic Use in a Single Intensive Care Unit
Brief Title: Effect of Copper Impregnated Textiles on Healthcare Associated Infections and Antibiotic Use
Status: Completed | Type: Observational
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Cupron Inc. (Industry)
Responsible Party: Principal Investigator, SShankaran, Assistant Professor, Internal Medicine, Division of Infectious Diseases, Eastern Virginia Medical School
Other Study IDs: 13-08-FB-0171
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Hospital Acquired Infection
Keywords: infection control; Prevention of hospital acquired infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Copper linens: One ward during each period (23 weeks each) used copper impregnated linen on the bed and as patient gowns. The second ward used regular linen on the bed and as patient gowns
  Interventions: Other: Copper impregnated linen

INTERVENTIONS:
Other: Copper impregnated linen — Copper impregnated linen was used in place of regular linen on one ward (out of two) for each period of the study. Each study period lasted for 23 weeks. After the washout period (3 weeks) the wards were switched.

SUMMARY:
This is a prospective Infection Control study comparing rates of antibiotic usage and infections in the General Intensive Care Unit (GICU) in beds with copper impregnated linens versus regular linens.

DETAILED DESCRIPTION:
One ward of the ICU had copper impregnated linen while the other had regular linen. This included sheets, pillowcases, towels and patient gowns. After the first 23 week period was completed, there was a 3 week washout period. After this, the wards were switched with the first using regular linen and the second using copper impregnated linen.

The investigators followed participants and documented any infections >48 hours after admission to the ICU. The number and days of antibiotics used for the infections were also documented. Using assigned study numbers, the investigators obtained demographic data: age, sex, co-morbid conditions, and admitting diagnosis. All participants were followed daily in the GICU and daily for 48 hours after transfer to the regular floor. Date of discharge will be obtained retrospectively. Infection control (IC) routinely obtains Methicillin Resistant Staphylococcus Aureus (MRSA) nasal swabs on all patients on admission to the GICU, once weekly while in GICU and then again on discharge from the GICU. They monitor the GICU patients for healthcare associated infections (HAI) that meet the National Healthcare Safety Network (NHSN) 146 definitions. The NHSN is a widely used HAI tracking system, and the infections documented included Ventilator associated pneumonia (VAP), Catheter related blood stream infections (CLABSI), catheter associate urinary tract infections (CAUTI) and Clostridium difficile associated diarrhea (CDAD). They also obtain information on decubitus ulcers (bed sores) that develop during hospital stay. Infection control also routinely monitors the isolation of multi-drug resistant bacteria, namely Vancomycin Resistant Enterococci (VRE), Extended Spectrum beta Lactamase producing organisms (ESBL) and Carbapenemase producing enterobacteriaceae (CRE) as well as Multi drug resistant (MDR ) Acinetobacter baumanii from cultures. This above information will be obtained from the IC nurses on a weekly basis by the investigators.

As most of the infections in the ICU do not meet strict NHSN criteria, the investigators defined an infection as: the physician diagnosing an infection, and then initiating antibiotics for the same.

Copper linen were implemented the same as regular linen. There was no difference in the nursing or physician staff on either side. No interventions were made other than existing hospital wide IC interventions

ELIGIBILITY:
Inclusion Criteria:All patients >18 years and <90 years who were admitted to the GICU during the study period

-

Exclusion Criteria:

1. Those that did not meet the age criteria as above.
2. Any patients with Menke's syndrome or Wilson's disease
3. Any patient with an allergy to copper or iodine
4. Any patient who wishes to opt out of participating

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years and <90 years who were admitted to the GICU during the study period
Sampling Method: Probability Sample
Enrollment: 1302 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Antibiotic usage in copper impregnated vs regular linen wards >48 hours after admission to ICU | Two study periods of 23 weeks each
  To assess whether the use of copper impregnated linens was associated with decreased use of antibiotics

SECONDARY OUTCOMES:
Decrease in clinical infection | Two study periods of 23 weeks each
  To assess whether the copper impregnated linen usage was associated with decrease in the number of clinical infections diagnosed by physicians
Decrease in NHSN infection | Two study periods of 23 weeks each
  Secondary measure included whether the copper impregnated linen usage was associated with decrease in the number of NHSN infections as defined by the infection control personnel

CONTACTS AND LOCATIONS:
Overall Officials: Shivanjali Shankaran, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Sentara Norfolk General Hospital, Norfolk, Virginia, United States

REFERENCES:
- [Background] Schmidt MG, Attaway Iii HH, Fairey SE, Steed LL, Michels HT, Salgado CD. Copper continuously limits the concentration of bacteria resident on bed rails within the intensive care unit. Infect Control Hosp Epidemiol. 2013 May;34(5):530-3. doi: 10.1086/670224. PMID 23571374
- [Background] Salgado CD, Sepkowitz KA, John JF, Cantey JR, Attaway HH, Freeman KD, Sharpe PA, Michels HT, Schmidt MG. Copper surfaces reduce the rate of healthcare-acquired infections in the intensive care unit. Infect Control Hosp Epidemiol. 2013 May;34(5):479-86. doi: 10.1086/670207. PMID 23571364
- [Background] Bilian X. Intrauterine devices. Best Pract Res Clin Obstet Gynaecol. 2002 Apr;16(2):155-68. doi: 10.1053/beog.2002.0267. PMID 12041959
- See also: NHSN infection definition — http://www.cdc.gov/nhsn/pdfs/pscmanual/17pscnosinfdef_current.pdf